CLINICAL TRIAL: NCT00466531
Title: A Phase I/IIa Trial For The Treatment of Relapsed or Chemotherapy Refractory Chronic Lymphocytic Leukemia or Indolent B Cell Lymphoma Using Autologous T Cells Genetically Targeted to the B Cell Specific Antigen CD19
Brief Title: Treatment of Relapsed or Chemotherapy Refractory Chronic Lymphocytic Leukemia or Indolent B Cell Lymphoma Using Autologous T Cells Genetically Targeted to the B Cell Specific Antigen CD19
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-138; MSKCC-06138
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; 06-138
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide

ARMS (1):
- Patients with CLL or indolent B-cell lymphoma (Experimental): The first stage is a standard 3-step phase I dose escalation trial to assess the safety of 19-28z CAR expressing autologous T cells with or without prior conditioning chemotherapy.Step 1, a cohort of pts will receive the lowest planned dose of 19-28z+ modified T cells. Step 2, a cohort of pts will receive cyclophosphamide conditioning chemotherapy followed by the lowest planned dose of 19-28z+ modified T cells. If less than 33% of pts in the cohort experience unanticipated dose-limiting toxicity,Step 3, a cohort of pts will be treated with the investigator's choice conditioning chemotherapy followed by the higher dose of 19-28z+ modified T cells. If less than 33% of pts in the initial cohort (Step 3) experience unanticipated dose-limiting toxicity, the cohort in Step 3 may be expanded to include up to 15 pts. In Step 3, an additional cohort of Waldenstrom's Macroglobulinemia (WM) pts will be treated with the investigator's choice conditioning chemotherapy followed by 19-28z+ T cells.
  Interventions: Biological: therapeutic autologous lymphocytes; Drug: cyclophosphamide

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Using T cells from the patient that have been treated in the laboratory may help the body build an effective immune response to kill cancer cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving laboratory-treated T cells together with cyclophosphamide may kill more cancer cells.

PURPOSE: This is a two-stage protocol, consisting of a single-institution phase I safety study and multi-institution phase IIa extension study.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase 1: The primary objective is to assess the safety of autologous T cells genetically modified to express chimeric antigen receptor (CAR) targeting CD19 antigen (19-28z) with or without conditioning chemotherapy.

• Phase IIa: The primary objective is to compare the relative engraftment and persistence of the two CAR modified CD19-targeted T cells expressing different co-stimulatory signaling domain CD28 (19-28z) and 4-1BB (CART-19:CD3z-4-1BB) in the CAR construct.

To compare the in vivo survival of genetically modified 19-28z CAR+ T cells after T cell infusion alone or in combination with conditioning chemotherapy.

* To compare the gene transfer/expression efficiency of the two viral vectors (retrovirus vs. lentivirus).
* To assess the anti-leukemic activity of adoptively transferred CD19-targeted modified T cells linked to the CD28 (19-28z) and 4-1BB signaling domains (CART-19:CD3z-4-1BB).

OUTLINE:

The first stage is a standard 3-step phase I dose escalation trial to assess the safety of 19-28z CAR expressing autologous T cells with or without prior conditioning chemotherapy. In Step 1, a cohort of patients will receive the lowest planned dose of 19-28z+ modified T cells. In Step 2, a cohort of patients will receive cyclophosphamide conditioning chemotherapy followed by the lowest planned dose of 19-28z+ modified T cells. If less than 33% of patients in the cohort (Step 2) experience unanticipated dose-limiting toxicity. In Step 3, a cohort of patients will be treated with the investigator's choice conditioning chemotherapy followed by the higher dose of 19-28z+ modified T cells. If less than 33% of patients in the initial cohort (Step 3) experience unanticipated dose-limiting toxicity, the cohort in Step 3 may be be expanded to include up to 15 patients. In Step 3, an additional cohort of Waldenstrom's Macroglobulinemia (WM) patients will be treated with the investigator's choice conditioning chemotherapy followed by 19-28z+ T cells. However, to maximize safety for WM patients, they will be treated at the lower dose of modified T cells (1x106 19-28z+ T cells/kg). If no toxicity is observed in the initial cohort, the dose may be increased in a standard 3-step dose-escalation scheme as described above.

In the Phase IIa extension part of the trial, 12 patients from MSKCC will be enrolled, and will be treated with co-infusion of 19-28z and CART-19:CD3z-4-1BB+ modified T cells mixed at 1:1 ratio at the MTD of T cells determined from the phase I trial.

ELIGIBILITY:
Inclusion:

• Patients must have the following CD19+ B cell leukemia or lymphoma either with relapsed or chemotherapy-refractory disease or with evidence of residual disease following therapy.

In all cases, patient's disease must be confirmed at MSKCC.

* CLL: Patients must have a diagnosis of CLL as evidenced by flow cytometry, bone marrow histology, and/or cytogenetics.
* Other low grade B-cell neoplasms are eligible for study, such as small lymphocytic lymphoma (SLL), follicular lymphoma, Waldenstrom's macroglobulinemia, hairy cell leukemia, marginal zone lymphomas, and mantle cell lymphomas.
* Creatinine ≤2.0 mg/100 ml, bilirubin ≤2.0 mg/100 ml, AST and ALT ≤3.0x normal, PT and PTT ≤ 2x normal outside the setting of stable chronic anticoagulation therapy, granulocytes ≥1,000/mm3, platelets ≥50,000/mm3, hemoglobin ≥8.0g/dl with transfusion support
* Adequate cardiac function (LVEF ≥40%) as assessed by ECHO or MUGA scan performed within 1 month of treatment.
* Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry.
* Life expectancy of > 3 months.

Exclusion:

* Karnofsky performance status <70.
* CLL patients with active transformed disease (Richter's transformation) are ineligible for enrollment on this study.
* Patients with following cardiac conditions will be excluded:
* New York Heart Association (NYHA) stage III or IV congestive heart failure
* Myocardial infarction ≤6 months prior to enrollment
* History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
* History of severe non-ischemic cardiomyopathy with EF ≤20%
* Patients with HIV, hepatitis B or hepatitis C infection are ineligible.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03-21; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety (phase I) | 1 year
efficacy of the two CD19-targeted T cell methods (phase II) | 1 year

SECONDARY OUTCOMES:
Antileukemic effect | 1 year
Comparison of in vivo survival of patients receiving genetically modified anti-CD19 T cells after T-cell infusion with vs without lymphodepleting therapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Brentjens RJ, Riviere I, Park JH, Davila ML, Wang X, Stefanski J, Taylor C, Yeh R, Bartido S, Borquez-Ojeda O, Olszewska M, Bernal Y, Pegram H, Przybylowski M, Hollyman D, Usachenko Y, Pirraglia D, Hosey J, Santos E, Halton E, Maslak P, Scheinberg D, Jurcic J, Heaney M, Heller G, Frattini M, Sadelain M. Safety and persistence of adoptively transferred autologous CD19-targeted T cells in patients with relapsed or chemotherapy refractory B-cell leukemias. Blood. 2011 Nov 3;118(18):4817-28. doi: 10.1182/blood-2011-04-348540. Epub 2011 Aug 17. PMID 21849486
- [Derived] Geyer MB, Riviere I, Senechal B, Wang X, Wang Y, Purdon TJ, Hsu M, Devlin SM, Palomba ML, Halton E, Bernal Y, van Leeuwen DG, Sadelain M, Park JH, Brentjens RJ. Safety and tolerability of conditioning chemotherapy followed by CD19-targeted CAR T cells for relapsed/refractory CLL. JCI Insight. 2019 Apr 2;5(9):e122627. doi: 10.1172/jci.insight.122627. PMID 30938714
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/